CLINICAL TRIAL: NCT05330026
Title: Ultrasound Imaging of the Diaphragm During Yoga Breathing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Teresa Emilia Fernandez Pardo, Principal investigator, Universidad Autonoma de Madrid
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CEI-120- 2409
Record Dates: First submitted 2022-02-04; First posted 2022-04-15 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Yoga
Keywords: breathing; diaphragm; ultrasound
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga practitioner (Experimental): The RUSI protocol for taking measurements with ultrasound for physiotherapists will be followed. Three measurements of each of the explorations will be made with the average of the three, pausing for 30 seconds between each repetition.
  Three variables will be analyzed: diaphragm thickness, its rate of contraction, and diaphragmatic excursion, all of them at rest, ujjayi breathing, and pursed-lip breathing.
  Interventions: Combination Product: Diaphragm´s study during yoga breathing
- Non yoga practitioner (Active Comparator): Each subject will have previously received (one week before taking the measurements) the instructions where the main researcher will have shown him what calm diaphragmatic breathing is like, as well as forced breathing at maximum inspired volume with neutral breathing, yoga breathing (ujjayi ) and pursed-lip breathing. During that week prior to taking measurements, the subjects should practice each breath for 20 minutes a day in order to have a good awareness of how to perform them correctly.
  The RUSI protocol for taking measurements with ultrasound for physiotherapists will be followed. Three measurements of each of the explorations will be made with the average of the three, pausing for 30 seconds between each repetition.
  Three variables will be analyzed: diaphragm thickness, its rate of contraction, and diaphragmatic excursion, all of them at rest, ujjayi breathing, and pursed-lip breathing.
  Interventions: Combination Product: Diaphragm´s study during yoga breathing

INTERVENTIONS:
Combination Product: Diaphragm´s study during yoga breathing — Study and compare the activation of the diaphragm during different breaths: rest, ujjayi and pursed lips

SUMMARY:
INTRODUCTION The practice of yoga in recent years is becoming more common. Originating in India, yoga combines physical postures with a philosophy of life and breathing (pranayama). One of the breaths used during yoga practice is the so-called ujjayi or victorious breath. It consists of the voluntary contraction of the muscles of the larynx both in inspiration and expiration. This reduces the diameter of the larynx, reducing airflow and thus increasing intrathoracic pressure, as well as increasing expiratory/inspiratory time and reducing respiratory rate and dead space. It also increases oxygen saturation in healthy subjects, increasing respiratory effort. Several studies have verified the relationship between ujjayi breathing and increased BRS (cardiovagal baroreflex sensitivity), by stimulation of the parasympathetic system at the glottis level.

This would favor a decrease in heart rate, as well as better control of stress and anxiety.

The cardiovascular and respiratory effects studied with ujjayi breathing have not evaluated the effect that this breath has on the activation of the respiratory muscles, mainly the diaphragm. The diaphragm is the main inspiratory muscle and as such, lung volumes and intrathoracic pressures created during respiration depend on its activation and position.

In recent years, ultrasound has become a technique widely used by pulmonologists and intensivists. It is an easy technique to perform, reproducible, non-ionizing, allows bilateral comparison, non-invasive and non-painful and whose results can broaden the information from other techniques such as spirometry and radiography.

There are standardized protocols to measure the diaphragmatic excursion, the thickness of the diaphragm HYPOTHESIS: ujjayi breathing is capable of generating greater activation of the diaphragm in subjects healthy with respect to spontaneous or pursed-lip breathing.

OBJECTIF: study and compare the activation and work of the diaphragm in different type of breathing (ujjayi, pursed lips and at rest) in healthy subjects who practice yoga or not. DESIGN: cross over study experimental, analytical and prospective. METHODOLOGY: 80 healthy subjets (40 yoga practitioners and 40 non yoga practitioners) participated at this study. All of them volunteers will undergo an ultrasound study of their diaphragm. To do this, following the stipulated protocol, three variables will be analyzed: diaphragm thickness, its rate of contraction, and diaphragmatic excursion, all of them at rest, ujjayi breathing, and pursed-lip breathing.

The ultrasound measurements will be taken by a single researcher, who is not the main one, and who will not know which group each of the subjects belongs to, thus avoiding an evaluation bias. To avoid bias and according to the RUSI regulations, the researcher will take 3 measurements of each of the explorations with the average of the 3.

ELIGIBILITY:
Inclusion Criteria:

* yoga practitioners for more than a year

Exclusion Criteria:

* respiratory pathology
* thoracic deformities
* neuromuscular diseases
* Under treatment with corticosteroids, muscle relaxants and/or barbiturates
* allergic episodes in the last 3 weeks
* thoracic or abdominal surgeries in the last 3 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Diaphragm thickness | Baseline, end maximal inspiration
  The assessment will be taken in the right hemidiaphragm since it is more accessible than the left through its hepatic window. To evaluate the thickness the investigators will use a linear probe at 10-12MHz, placing it perpendicular to the intercostal space between the 9th and 10th rib, in the anterior part of the axillary line.
  At this level, 3 parallel layers with different echogenicity corresponding to the pleura, diaphragm and peritoneum will be observed. The distance between the inner edge of the pleural line and the inner edge of the peritoneal line will be measured.

SECONDARY OUTCOMES:
Diaphragm excursion | Baseline, end maximal inspiration
  The distance it makes in inspiration will be measured, when it contracts and descends. A 2.5 to 3.5 MHz convex probe will be used.
  The probe will be positioned firmly below the right costal arch and on the line corresponding to the middle of the clavicle, orienting it cranially. The investigators will visualize the dome of the right hemidiaphragm that appears as a thick hyperechoic line. The investigators look for the highest diaphragmatic position, which is the part of the diaphragm that produces the greatest cranial-caudal excursion. The M mode modality will be activated, which provides us with the pattern of diaphragmatic movement.
  It will be measured from the highest point of the diaphragmatic dome (end expiration, in functional residual capacity) to the lowest point achieved at the end of each inspiration.
Activation speed | Baseline, end maximal inspiration
  It is an indirect measurement that is calculated by dividing the diaphragm amplitude in cm by the inspiratory time in seconds. Will be measured with TM mode

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Autónoma de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
All the researchers will participate in all the study phases